CLINICAL TRIAL: NCT06940570
Title: A Randomized Single Center Trial to Determine the Efficacy of Methadone as a First Line Agent in the Reduction and Treatment of Pain in Pediatric Patients Undergoing Hematopoietic Stem Cell Transplantation
Brief Title: Methadone as an Alternative Treatment for Children Underdoing HSCT
Acronym: MATCH
Status: Suspended | Phase: Phase 3 | Type: Interventional
Why Stopped: Study is closed with the IRB due to no funding. May resume once funding is obtained.
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, James DeMasi, Nurse Practitioner - Anesthesiology and Pain Management, Children's Health
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: STU-2022-0876
Record Dates: First submitted 2025-03-17; First posted 2025-04-23 (Actual); Last update posted 2025-10-23 (Actual); Status verified 2025-10

CONDITIONS: Leukemia; Aplastic Anemia; Bone Marrow Failure Syndromes; SCID
Keywords: intractable pain; methadone; mucositis; pediatric cancer; hematopoietic stem cell transplantation
MeSH Terms: conditions — Leukemia; Anemia, Aplastic; Bone Marrow Failure Disorders; Pain, Intractable; Mucositis; Neoplasms | interventions — Passive Cutaneous Anaphylaxis; Methadone; Morphine; Hydromorphone

STUDY DESIGN:
Intervention Model Description: This will be a randomized control study where pt is placed in one of two groups, methadone receiving plus PCA push only (experimental) OR PCA/continuous infusion without methadone (control)
Who Masked: Participant, Care Provider
Masking Description: Parent would be masked as well
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group A: Control Arm (n = 30) (Active Comparator): Pt will receive: PCA opioid will include morphine OR hydromorphone (if patient has a sensitivity or is unable to tolerate or allergic to morphine). This is the exclusive medication/opioid in this arm. The starting doses will be as follows:
  * Starting dose for basal infusion of morphine is 0.02 mg/kg/hour up to a maximum of 50 kg.
  * Starting PCA dose for morphine is 0.02 mg/kg every 15 minutes for a lockout of 0.1 mg/kg up to a maximum of 50 kg or ideal body weight (PCA starting dose should be no more than 1 mg/push and no more than 5 mg/hour lockout).
  * Starting dose for basal infusion of hydromorphone is 0.003 mg/kg/hour up to a maximum of 50 kg IBW.
  * Starting PCA dose for hydromorphone is 0.003 mg/kg every 15 minutes for an hourly maximum lockout of 0.012 mg/kg up to a maximum of 50 kg (PCA start
  * PCA medications may be titrated up or down by 20-50% each day for desired analgesic effect with improved pain score, continue to engraftment or when medicine is no longer needed.
  Interventions: Drug: PCA Alone (SOC)
- Group B: Study or Experimental Arm (n = 30) (Experimental): The second arm will be methadone therapy that is scheduled to be given every 8 hours in addition to an on demand PCA. On demand PCA dosing will be the same as control arm but with NO basal/continuous rate. Intravenous methadone will be replacing basal infusion and serve as basal drug in place of continuous medication.
  * Starting dose for intravenous methadone is 0.1 mg/kg IV Q8hr up to a maximum of 50 kg. Singular starting methadone will be maximum of 5 mg.
  * Methadone may be increased by 20-50% every 48 hours due to half-life of medication. Reduction in analgesia will need to be monitored daily following a change. However, additional methadone increase should not occur until 48 hours have passed to allow for steady state of new dose to take effect. Reduction of methadone dosing by 20-50% can be made anytime per discretion of provider or if concerned about an adverse effect from the methadone.
  This will continue until engraftment or until medicine is no longer needed.
  Interventions: Drug: PCA plus methadone (Experimental)

INTERVENTIONS:
Drug: PCA plus methadone (Experimental) — This study is novel. There are no other interventions to distinguish in this or another study.
  Other Names: Addition of methadone to standard of care (SOC)
  Arms: Group B: Study or Experimental Arm (n = 30)
Drug: PCA Alone (SOC) — PCA Alone (Control) arm. PCA opioid will include morphine OR hydromorphone (if patient has a sensitivity or is unable to tolerate or allergic to morphine).
  Other Names: Morphine OR Hydromorphone
  Arms: Group A: Control Arm (n = 30)

SUMMARY:
Mucositis is a normal side effect of stem cell transplant which happens as a result of chemotherapy being given prior to a new donor cell infusion (bone marrow transplant). The chemotherapy will kill cancer cells, but good cells, such as those in the mouth, are killed too. The mouth cells going away causes the areas in the mouth to be blistered, irritated, sore, and extremely painful. Pain medication (usually morphine or hydromorphone if allergic to morphine) are given when oral blisters are seen or felt by patient in patient's mouth. However, one pain medication given through a vein in the patient may or may not be effective and providers are often challenged with providing good pain control while waiting for the new donor cells to grow, which will then heal the mouth. This is a period of waiting that is 6-8 weeks.

The investigators know that methadone, a second pain medication, may decrease pain in a different way than morphine. This is because methadone works in a different way in the brain than morphine. By giving these pain medicines together, the hope of the study is to show decreased pain while waiting for new cells to grow.

The goal of this clinical trial is to hope to learn whether adding methadone (second pain medication) to the current pain medication which is morphine alone (all patients will receive this pain medication) will help reduce the pain experience of participant. Current treatment of morphine alone is sometimes not entirely effective and so any improvement of pain while waiting for new cells to grow is one of the goals of this study. If methadone is effective in decreasing pain, then patients may benefit in the future from using these two medications up front when getting a transplant.

Participant in this study between 6-18 years of age and is needing a stem cell transplant for a disease that can potentially be cured by transplantation.

Participant in this study is receiving chemotherapy and/or radiation conditioning that can cause mucositis. Participants are being asked to participate in this study because participants meet criteria to receive methadone that may or may not reduce pain experience versus just being given morphine alone, which is what all patients are given when the participants have mucositis.

The main goal of the study is to see if less opioid (pain medication) when methadone is added in comparison to participant who uses PCA only. The investigators also want to learn if patient's overall function is improved if given methadone. Another goal would be to see the number of TPN days the participant received and if the participant who was given methadone began to eat sooner. Other smaller goals include learning about side effects of methadone, and if the hospital stay is less for those who receive the study medication.

This medication will be given at Children's Medical Center of Dallas while participant is admitted for the stem cell transplant. There is no sponsor that is funding the study and this drug will be given free of charge in exchange for participation in the study

DETAILED DESCRIPTION:
Given high reports of pain while despite receiving PCA during transplant, our current management of mucositis induced pain is suboptimal. In a study of children receiving transplantation, pain was a main concern for this cohort during and after transplantation. The investigators propose to conduct this study to determine if methadone used as a primary analgesic in patients with mucositis can improve the current standard of care which will be demonstrated by improved pain scores, maintenance of functionality, and recovery during and following HSCT. This study will be a single blind randomized controlled design. Patients will be randomly assigned by permuted block randomization in groups of eight. Patient will be randomly assigned to receive either basal/PCA of one opioid (control) in the first arm OR PCA plus methadone where methadone will be used as basal long-acting medication (experimental).

Study subjects will be children who are undergoing an autologous or allogeneic stem cell transplant receiving a myeloablative regimen and meet all inclusion criteria. This unique population is being studied as it is a controlled setting where the PI can anticipate pain in >90% of the patients following ablation, the number of patients who experience mucositis after receiving ablative conditioning. The study will only be conducted in the inpatient stem cell transplant setting and no follow up should be necessary when these subjects are discharged from the hospital after transplant.

The following goals of the study are as follows:

1. Will the concomitant administration of intravenous administered methadone with on demand opioid PCA improve pain score numbers in the PCA/methadone arm (experimental) in comparison to a continuous infusion PCA with demand opioid arm (control, standard of care)?
2. Will the administration of methadone with increased individualized titration result in a reduction of 25% in total morphine milligram equivalents (MME) in experimental versus control arm?
3. Will the methadone experimental arm increase functionality during transplantation period?
4. Will those receiving methadone have reduced TPN days during hospital stay as compared to control arm?
5. Will the child resumes oral intake more rapidly compared to control arm?
6. The investigators also want to describe adverse events and incidence associated with methadone when administered in combination with morphine or hydromorphone, specifically QTc prolongation that has been documented with study medication.

ELIGIBILITY:
Inclusion Criteria:

* All subjects admitted will receive a myeloablative conditioning regimen followed by autologous or allogeneic bone marrow transplant during transplant admission. Conditioning may include chemotherapy, radiation, or a combination of both methods to be determined by primary attending transplant physician. Diagnoses will include but not limited to those with liquid tumors, solid tumors, hematological/congenital blood disorders, or severe combined immunodeficiency syndromes.
* Subjects must be 6-18 years of age and demonstrate understanding of PCA use or have a parent available for PCA by proxy, meaning parent can push the button for the patient. Patient maximum age is 18 years old. PCA proxy in compliance with Pain Assessment and Management policy per institution.
* Performance status: Karnofsky/Lansky >50% prior to receiving conditioning.
* Be cognitively able to utilize and understand patient-controlled analgesia (PCA).
* Informed consent will be obtained from all participants or their parents or guardians, assent will be obtained from children ages 10-17 years of age per institutional policy.

Exclusion Criteria:

* QT prolongation prior to receiving myeloablative conditioning as evidenced by QTc being >450 for both girls and boys prior to starting methadone.
* Medical history of QT prolongation, VF, or VT.
* Patients on chronic pain medications on admission or have received more than 30 days of continuous opioids over the past month.
* Patients receiving a non-myeloablative regimen or no conditioning.
* Neurological or psychiatric condition that could confound reliable assessment of pain and sedation (non-verbal, global delay).
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to morphine or other agents used in study.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that, in the opinion of the investigator, would limit compliance with study requirements.
* History of opioid misuse disorder OR opioid risk assessment tool score >8.

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 60 (Estimated)
Dates: Start 2028-01-01 (Estimated); Primary Completion 2029-08 (Estimated); Study Completion 2029-08-01 (Estimated)

PRIMARY OUTCOMES:
Reduction of pain score | Daily after completion of conditioning (day +7 to day +14) through discharge (approximately day +60)
  The purpose of the study is to compare methadone versus standard of care at this center of morphine/hydromorphone PCA and see if methadone is superior to the standard of care as evidenced by reduction in pain scores during inpatient transplant.
  To determine whether concomitant administration of intravenous administered methadone with on demand opioid PCA will improve pain score numbers in the PCA/methadone arm by 25% in comparison to a continuous infusion PCA with demand opioid arm.

SECONDARY OUTCOMES:
REDUCTION OF OPIOID RECEIVED as evidenced by 25% reduction of MME in experimental arm in comparison to control arm | Daily after completion of conditioning (day +7 to day +14) through discharge (approximately day +60)
  To determine if methadone (starting dose of 0.1 mg/kg IV Q8hr) with increased titration will result in a reduction of 25% in total morphine milligram equivalents (MME) per day in children who have mucositis following ablative conditioning and subsequent allogeneic or autologous HSCT
IMPROVEMENT OF FUNCTIONALITY as evidenced by higher functionality scores in experimental arm in comparison to control | Day 0 (stem cell infusion)
  To determine how administration of methadone affects functionality during transplantation period
REDUCED NUMBER OF DAYS ON PARENTERAL NUTRITION as evidenced by reduced number of TPN days in experimental arm in comparison to control | From enrollment (initiation of TPN- typically on day +1) to engraftment day AND date when able to take solid food again (day just prior to discharge-approx. day+50 to day+60)
  To determine if the overall TPN days are reduced during hospital stay in experimental arm as compared to the standard PCA regimen
INCREASED RETURN TO ORAL LIQUID INTAKE as evidenced by more rapid return to tolerating clears in experimental group versus control | From enrollment (initiation of TPN- typically on day +1) to engraftment day AND date when able to take solid food again (day just prior to discharge-approx. day+50 to day+60)
  To determine if child resumes oral intake more rapidly compared to control arm
Adverse events | From first dose of methadone administered (day +1- day +7) until prior to discharge (approximately day +60)
  To describe adverse events and incidence associated with methadone when administered in combination with morphine or hydromorphone, specifically QTc prolongation that has been documented with study medication

CONTACTS AND LOCATIONS:
Overall Officials: Victor M Aquino, MD, Principal Investigator — UT Southwestern Department of Pediatric Oncology and Stem Cell Transplant
Locations (1):
- Children's Health of Dallas, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No
There is no reason to share individualized participant data in this study. My plan is to deidentify all data and all data will be anonymous.

REFERENCES:
- [Background] Portenoy RK. Treatment of cancer pain. Lancet. 2011 Jun 25;377(9784):2236-47. doi: 10.1016/S0140-6736(11)60236-5. PMID 21704873
- [Background] Jacob E. Neuropathic pain in children with cancer. J Pediatr Oncol Nurs. 2004 Nov-Dec;21(6):350-7. doi: 10.1177/1043454204270251. PMID 15475472
- [Background] Habashy C, Springer E, Hall EA, Anghelescu DL. Methadone for Pain Management in Children with Cancer. Paediatr Drugs. 2018 Oct;20(5):409-416. doi: 10.1007/s40272-018-0304-2. PMID 30047027
- [Background] Vasquenza K, Ruble K, Chen A, Billett C, Kozlowski L, Atwater S, Kost-Byerly S. Pain Management for Children during Bone Marrow and Stem Cell Transplantation. Pain Manag Nurs. 2015 Jun;16(3):156-62. doi: 10.1016/j.pmn.2014.05.005. Epub 2014 Sep 26. PMID 25267531
- [Background] White MC, Hommers C, Parry S, Stoddart PA. Pain management in 100 episodes of severe mucositis in children. Paediatr Anaesth. 2011 Apr;21(4):411-6. doi: 10.1111/j.1460-9592.2010.03515.x. Epub 2011 Jan 21. PMID 21251145
- [Background] Varni JW, Burwinkle TM, Katz ER, Meeske K, Dickinson P. The PedsQL in pediatric cancer: reliability and validity of the Pediatric Quality of Life Inventory Generic Core Scales, Multidimensional Fatigue Scale, and Cancer Module. Cancer. 2002 Apr 1;94(7):2090-106. doi: 10.1002/cncr.10428. PMID 11932914
- [Background] Vagliano L, Feraut C, Gobetto G, Trunfio A, Errico A, Campani V, Costazza G, Mega A, Matozzo V, Berni M, Alberani F, Banfi MM, Martinelli L, Munaron S, Orlando L, Lubiato L, Leanza S, Guerrato R, Rossetti A, Messina M, Barzetti L, Satta G, Dimonte V. Incidence and severity of oral mucositis in patients undergoing haematopoietic SCT--results of a multicentre study. Bone Marrow Transplant. 2011 May;46(5):727-32. doi: 10.1038/bmt.2010.184. Epub 2010 Sep 6. PMID 20818449
- [Background] Tomlinson D, Judd P, Hendershot E, Maloney AM, Sung L. Measurement of oral mucositis in children: a review of the literature. Support Care Cancer. 2007 Nov;15(11):1251-1258. doi: 10.1007/s00520-007-0323-y. Epub 2007 Aug 28. PMID 17724620
- [Background] Sonis ST, Elting LS, Keefe D, Peterson DE, Schubert M, Hauer-Jensen M, Bekele BN, Raber-Durlacher J, Donnelly JP, Rubenstein EB; Mucositis Study Section of the Multinational Association for Supportive Care in Cancer; International Society for Oral Oncology. Perspectives on cancer therapy-induced mucosal injury: pathogenesis, measurement, epidemiology, and consequences for patients. Cancer. 2004 May 1;100(9 Suppl):1995-2025. doi: 10.1002/cncr.20162. PMID 15108222
- [Background] Sonis ST. The pathobiology of mucositis. Nat Rev Cancer. 2004 Apr;4(4):277-84. doi: 10.1038/nrc1318. No abstract available. PMID 15057287
- [Background] Sirkia K, Hovi L, Pouttu J, Saarinen-Pihkala UM. Pain medication during terminal care of children with cancer. J Pain Symptom Manage. 1998 Apr;15(4):220-6. doi: 10.1016/s0885-3924(98)00366-2. PMID 9601156
- [Background] Scully C, Sonis S, Diz PD. Oral mucositis. Oral Dis. 2006 May;12(3):229-41. doi: 10.1111/j.1601-0825.2006.01258.x. PMID 16700732
- [Background] Schiessl C, Gravou C, Zernikow B, Sittl R, Griessinger N. Use of patient-controlled analgesia for pain control in dying children. Support Care Cancer. 2008 May;16(5):531-6. doi: 10.1007/s00520-008-0408-2. Epub 2008 Feb 15. PMID 18274785
- [Background] Rose-Ped AM, Bellm LA, Epstein JB, Trotti A, Gwede C, Fuchs HJ. Complications of radiation therapy for head and neck cancers. The patient's perspective. Cancer Nurs. 2002 Dec;25(6):461-7; quiz 468-9. doi: 10.1097/00002820-200212000-00010. PMID 12464838
- [Background] Pearson EC, Woosley RL. QT prolongation and torsades de pointes among methadone users: reports to the FDA spontaneous reporting system. Pharmacoepidemiol Drug Saf. 2005 Nov;14(11):747-53. doi: 10.1002/pds.1112. PMID 15918160
- [Background] Parsons HA, de la Cruz M, El Osta B, Li Z, Calderon B, Palmer JL, Bruera E. Methadone initiation and rotation in the outpatient setting for patients with cancer pain. Cancer. 2010 Jan 15;116(2):520-8. doi: 10.1002/cncr.24754. PMID 19924788
- [Background] Papas AS, Clark RE, Martuscelli G, O'Loughlin KT, Johansen E, Miller KB. A prospective, randomized trial for the prevention of mucositis in patients undergoing hematopoietic stem cell transplantation. Bone Marrow Transplant. 2003 Apr;31(8):705-12. doi: 10.1038/sj.bmt.1703870. PMID 12692611
- [Background] Moulin DE, Clark AJ, Gilron I, Ware MA, Watson CP, Sessle BJ, Coderre T, Morley-Forster PK, Stinson J, Boulanger A, Peng P, Finley GA, Taenzer P, Squire P, Dion D, Cholkan A, Gilani A, Gordon A, Henry J, Jovey R, Lynch M, Mailis-Gagnon A, Panju A, Rollman GB, Velly A; Canadian Pain Society. Pharmacological management of chronic neuropathic pain - consensus statement and guidelines from the Canadian Pain Society. Pain Res Manag. 2007 Spring;12(1):13-21. doi: 10.1155/2007/730785. PMID 17372630
- [Background] Mercadante S. Methadone in cancer pain. Eur J Pain. 1997;1(2):77-83; discussion 84-5. doi: 10.1016/s1090-3801(97)90064-1. PMID 15102407
- [Background] Mercadante S, Porzio G, Ferrera P, Fulfaro F, Aielli F, Verna L, Villari P, Ficorella C, Gebbia V, Riina S, Casuccio A, Mangione S. Sustained-release oral morphine versus transdermal fentanyl and oral methadone in cancer pain management. Eur J Pain. 2008 Nov;12(8):1040-6. doi: 10.1016/j.ejpain.2008.01.013. Epub 2008 Mar 18. PMID 18353696
- [Background] Mercadante S, Bruera E. Opioid switching in cancer pain: From the beginning to nowadays. Crit Rev Oncol Hematol. 2016 Mar;99:241-8. doi: 10.1016/j.critrevonc.2015.12.011. Epub 2015 Dec 29. PMID 26806145
- [Background] McNicol ED, Ferguson MC, Hudcova J. Patient controlled opioid analgesia versus non-patient controlled opioid analgesia for postoperative pain. Cochrane Database Syst Rev. 2015 Jun 2;2015(6):CD003348. doi: 10.1002/14651858.CD003348.pub3. PMID 26035341
- [Background] Madden K, Liu D, Bruera E. Attitudes, Beliefs, and Practices of Pediatric Palliative Care Physicians Regarding the Use of Methadone in Children With Advanced Cancer. J Pain Symptom Manage. 2019 Feb;57(2):260-265. doi: 10.1016/j.jpainsymman.2018.11.009. Epub 2018 Nov 15. PMID 30447383
- [Background] Lawitschka A, Guclu ED, Varni JW, Putz M, Wolff D, Pavletic S, Greinix H, Peters C, Felder-Puig R. Health-related quality of life in pediatric patients after allogeneic SCT: development of the PedsQL Stem Cell Transplant module and results of a pilot study. Bone Marrow Transplant. 2014 Aug;49(8):1093-7. doi: 10.1038/bmt.2014.96. Epub 2014 May 12. PMID 24820217
- [Background] Kao DP, Haigney MC, Mehler PS, Krantz MJ. Arrhythmia associated with buprenorphine and methadone reported to the Food and Drug Administration. Addiction. 2015 Sep;110(9):1468-75. doi: 10.1111/add.13013. PMID 26075588
- [Background] Gupta A, Lawrence AT, Krishnan K, Kavinsky CJ, Trohman RG. Current concepts in the mechanisms and management of drug-induced QT prolongation and torsade de pointes. Am Heart J. 2007 Jun;153(6):891-9. doi: 10.1016/j.ahj.2007.01.040. PMID 17540188
- [Background] Gorman AL, Elliott KJ, Inturrisi CE. The d- and l-isomers of methadone bind to the non-competitive site on the N-methyl-D-aspartate (NMDA) receptor in rat forebrain and spinal cord. Neurosci Lett. 1997 Feb 14;223(1):5-8. doi: 10.1016/s0304-3940(97)13391-2. PMID 9058409
- [Background] Glotzbecker B, Duncan C, Alyea E 3rd, Campbell B, Soiffer R. Important drug interactions in hematopoietic stem cell transplantation: what every physician should know. Biol Blood Marrow Transplant. 2012 Jul;18(7):989-1006. doi: 10.1016/j.bbmt.2011.11.029. Epub 2011 Dec 7. PMID 22155504
- [Background] Gai N, Naser B, Hanley J, Peliowski A, Hayes J, Aoyama K. A practical guide to acute pain management in children. J Anesth. 2020 Jun;34(3):421-433. doi: 10.1007/s00540-020-02767-x. Epub 2020 Mar 31. PMID 32236681
- [Background] Ehrentraut JH, Kern KD, Long SA, An AQ, Faughnan LG, Anghelescu DL. Opioid misuse behaviors in adolescents and young adults in a hematology/oncology setting. J Pediatr Psychol. 2014 Nov-Dec;39(10):1149-60. doi: 10.1093/jpepsy/jsu072. Epub 2014 Sep 14. PMID 25225182
- [Background] Cravero JP, Agarwal R, Berde C, Birmingham P, Cote CJ, Galinkin J, Isaac L, Kost-Byerly S, Krodel D, Maxwell L, Voepel-Lewis T, Sethna N, Wilder R. The Society for Pediatric Anesthesia recommendations for the use of opioids in children during the perioperative period. Paediatr Anaesth. 2019 Jun;29(6):547-571. doi: 10.1111/pan.13639. Epub 2019 Jun 11. PMID 30929307
- [Background] Bruera E, Palmer JL, Bosnjak S, Rico MA, Moyano J, Sweeney C, Strasser F, Willey J, Bertolino M, Mathias C, Spruyt O, Fisch MJ. Methadone versus morphine as a first-line strong opioid for cancer pain: a randomized, double-blind study. J Clin Oncol. 2004 Jan 1;22(1):185-92. doi: 10.1200/JCO.2004.03.172. PMID 14701781
- [Background] Codd EE, Shank RP, Schupsky JJ, Raffa RB. Serotonin and norepinephrine uptake inhibiting activity of centrally acting analgesics: structural determinants and role in antinociception. J Pharmacol Exp Ther. 1995 Sep;274(3):1263-70. PMID 7562497
- [Background] CDC morphine to methadone mg eq conversion data accessed on June 19, 2020 at https://www.cdc.gov/drugoverdose/pdf/calculating_total_daily_dose-a.pdf
- [Background] Boisvert-Plante V, Poulin-Harnois C, Ingelmo P, Einhorn LM. What we know and what we don't know about the perioperative use of methadone in children and adolescents. Paediatr Anaesth. 2023 Mar;33(3):185-192. doi: 10.1111/pan.14584. Epub 2022 Nov 11. PMID 36281540
- [Background] Blijlevens NM, Donnelly JP, De Pauw BE. Mucosal barrier injury: biology, pathology, clinical counterparts and consequences of intensive treatment for haematological malignancy: an overview. Bone Marrow Transplant. 2000 Jun;25(12):1269-78. doi: 10.1038/sj.bmt.1702447. PMID 10871732
- [Background] Barker CC, Anderson RA, Sauve RS, Butzner JD. GI complications in pediatric patients post-BMT. Bone Marrow Transplant. 2005 Jul;36(1):51-8. doi: 10.1038/sj.bmt.1705004. PMID 15908980
- [Background] Anghelescu DL, Oakes L, Popenhagen M. Management of cancer pain in neonates, children and adolescents. In: de Leon-Casasola, OA., editor. Cancer Pain: Pharmacological, Interventional, and Palliative Care Approaches. 1st ed., Philadelphia: Saunders Elsevier; 2006. P 509-521
- [Background] American Society of Anesthesiologists Task Force on Acute Pain Management. Practice guidelines for acute pain management in the perioperative setting: an updated report by the American Society of Anesthesiologists Task Force on Acute Pain Management. Anesthesiology. 2012 Feb;116(2):248-73. doi: 10.1097/ALN.0b013e31823c1030. No abstract available. PMID 22227789